CLINICAL TRIAL: NCT03750344
Title: ChroniSense Polso Wrist Worn Respiration Rate Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChroniSense Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR 2018-305
Record Dates: First submitted 2018-11-18; First posted 2018-11-23 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2018-11

CONDITIONS: Respiratory Rate
Keywords: Respiratory Rate
MeSH Terms: interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- ChroniSense Polso Respiratory Rate (Experimental)
  Interventions: Device: Diagnostic test

INTERVENTIONS:
Device: Diagnostic test — Comparison of respiratory rates in normal subjects as observational with end tidal CO2. No treatment or interventions will be performed

SUMMARY:
20 volunteer test subjects will be entered into an accuracy study that is designed to validate accuracy of the respiratory rate of the Polso Monitoring system

DETAILED DESCRIPTION:
20 volunteer test subjects will be entered into an accuracy study that is designed to validate accuracy of the respiratory rate of the Polso Monitoring system.

A range of stable respiratory rates will be elicited from each volunteer test subject. The rates will be approximately 5, 10, 15, 20, 25, 30, 35, 40 and 45 breaths per minute; with some natural variation from these exact numbers.

Each subject will be instrumented with an open system mask that allows for measurement of the end tidal carbon dioxide (EtCO2) respiratory rate and tidal volume. The EtCO2 monitor will be used as the Accuracy Reference Device (Reference) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject is adult over 18 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker
* Male or female of any race
* Wrist circumference with the range of 5.5-8 inches (13 to 21cm)

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. Tattoo in the optical path which would limit the ability to test sites needed for the study.
* Subjects with known respiratory conditions such as:

  * uncontrolled / severe asthma,
  * flu,
  * pneumonia / bronchitis,
  * shortness of breath / respiratory distress,
  * respiratory or lung surgery,
  * emphysema, COPD, lung disease
* Subjects with self-reported heart or cardiovascular conditions such as:

  * have had cardiovascular surgery
  * Chest pain (angina)
  * heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia
  * previous heart attack
  * blocked artery
  * unexplained shortness of breath
  * congestive heart failure (CHF)
  * history of stroke
  * transient ischemic attack
  * carotid artery disease
  * myocardial ischemia
  * myocardial infarction
  * cardiomyopathy
* Self-reported health conditions as identified in the Health Assessment Form

  * diabetes,
  * uncontrolled thyroid disease,
  * kidney disease / chronic renal impairment,
  * history of seizures (except childhood febrile seizures),
  * epilepsy,
  * history of unexplained syncope,
  * recent history of frequent migraine headaches,
  * recent head injury within the last 2 months,
* Cancer / chemotherapy
* Other known health condition should be considered upon disclosure in health assessment form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate Accuracy of Polso Monitoring System | Through study completion, 1 month average
  Respiratory Rate of test subject as compared to CO2 of End Tidal Carbon. Twenty second periods will be averaged to provide one respiratory rate value. Each stable respiratory rate plateau will result in four of these respiratory rate values which will be included in the ARMS calculation. The endpoint of interest is accuracy as measured by the Accuracy root-mean-square (Arms) difference between the device under test (DUT) and the reference respiratory rate system (Ref) for all stable respiratory periods. Acceptance criteria ARMS <3

CONTACTS AND LOCATIONS:
Overall Officials: Arthur D Cabrera, MD, Study Director — Avista Adventist Hospital
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No